CLINICAL TRIAL: NCT06170931
Title: Comparison Of Outcomes After Bilateral Simultaneous Total Knee Arthroplasty Using Posterior-Substituting Versus Cruciate-Retaining Prostheses
Brief Title: Comparison Of Outcomes After Knee Arthroplasty Using Posterior-Substituting Versus Cruciate-Retaining Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00013890
Record Dates: First submitted 2023-11-20; First posted 2023-12-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Total Knee Arthroplasty
Keywords: Knee; total knee arthroplasty; posterior cruciate ligament-substituting; posterior cruciate ligament-retaining

STUDY DESIGN:
Intervention Model Description: Patients with the same stage of knee osteoarthritis in both knees were selected. Total knee arthroplasty was performed in the same session by making the appropriate design for the appropriate knee simultaneously. Preoperative and postoperative joint range of motion examinations were performed on both knees separately. WOMAC and OXFORD scores were examined separately for both knees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A knee of a patient with osteoarthritis of both knees (Active Comparator): Posterior cruciate ligament protective approach in patients with knee osteoarthritis
  Interventions: Procedure: posterior cruciate ligament-retaining prostheses
- The other knee of a patient with osteoarthritis in both knees (Active Comparator): Posterior cruciate ligament transection approach in patients with knee osteoarthritis
  Interventions: Procedure: posterior cruciate ligament-substituting prostheses

INTERVENTIONS:
Procedure: posterior cruciate ligament-retaining prostheses — Posterior cruciate ligament protective approach in patients with knee osteoarthritis
  Arms: A knee of a patient with osteoarthritis of both knees
Procedure: posterior cruciate ligament-substituting prostheses — Posterior cruciate ligament transection approach in patients with knee osteoarthritis
  Arms: The other knee of a patient with osteoarthritis in both knees

SUMMARY:
Total knee replacement is used in the treatment of patients with knee arthritis, rheumatoid arthritis and other knee disorders. Today, there are basically two designs; It cuts the posterior cruciate ligament (PS) and protects the posterior cruciate ligament (CR). Although there is no clear study suggesting which design is better, research on this subject has increased recently. the investigators aim is to define the superiority of these two designs over each other. Preoperative and postoperative joint range of motion examinations were performed on both knees separately. WOMAC and OXFORD scores were examined separately for both knees.

DETAILED DESCRIPTION:
Total knee arthroplasty is used to treat patients with osteoarthritis, rheumatoid arthritis, and other knee disorders. Today, there are basically two primary designs; posterior cruciate Substituting (PS) and protects the posterior cruciate -Retaining (CR). However, it is still controversial which approach is good, as both CR and PS have advantages and disadvantages. Proponents of the posterior cruciate retaining system argue that it provides natural stability, wider joint range of motion, better proprioception, and better knee kinematics. In addition, proponents of the posterior cruciate substituting system argue that it provides more harmonious articulation and a wider flexion range.

As a result, although there is no clear study suggesting which design is better, research on this subject has increased recently. Our aim is to define the superiority of these two designs over each other.

Patients with the same stage of knee osteoarthritis in both knees were selected. Total knee arthroplasty was performed in the same session by making the appropriate design for the appropriate knee simultaneously. Preoperative and postoperative joint range of motion examinations were performed on both knees separately. WOMAC and OXFORD scores were examined separately for both knees.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary osteoarthritis of both knees
2. Patients with secondary osteoarthritis of both knees

Exclusion Criteria:

1. Patients with primary osteoarthritis in both knees and undergoing unilateral knee prosthesis
2. Patients with secondary osteoarthritis in both knees and who underwent unilateral knee prosthesis
3. Patients with primary osteoarthritis in both knees and who underwent bilateral knee prosthesis in different sessions
4. Patients with secondary osteoarthritis in both knees and who underwent bilateral knee prosthetics in different sessions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Range of motions | 3 year
  Preoperative and postoperative knee flexion and extension degrees of the patients were measured.

SECONDARY OUTCOMES:
WOMAC Score (Score from 0 to 100) | 3 year
  Preoperative and postoperative WOMAC score of the patients were examined.
OXFORD Knee Score(Score from 0 to 60) | 3 year
  Preoperative and postoperative OXFORD score of the patients were examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not think it is right that the data of the patients in the study can be seen by everyone.

REFERENCES:
- [Background] Li N, Tan Y, Deng Y, Chen L. Posterior cruciate-retaining versus posterior stabilized total knee arthroplasty: a meta-analysis of randomized controlled trials. Knee Surg Sports Traumatol Arthrosc. 2014 Mar;22(3):556-64. doi: 10.1007/s00167-012-2275-0. Epub 2012 Nov 3. PMID 23117166
- [Background] Rossi R, Bruzzone M, Bonasia DE, Marmotti A, Castoldi F. Evaluation of tibial rotational alignment in total knee arthroplasty: a cadaver study. Knee Surg Sports Traumatol Arthrosc. 2010 Jul;18(7):889-93. doi: 10.1007/s00167-009-1023-6. Epub 2010 Jan 8. PMID 20057997
- [Background] Insall JN, Lachiewicz PF, Burstein AH. The posterior stabilized condylar prosthesis: a modification of the total condylar design. Two to four-year clinical experience. J Bone Joint Surg Am. 1982 Dec;64(9):1317-23. No abstract available. PMID 7142239
- [Background] In Y, Kim JM, Woo YK, Choi NY, Sohn JM, Koh HS. Factors affecting flexion gap tightness in cruciate-retaining total knee arthroplasty. J Arthroplasty. 2009 Feb;24(2):317-21. doi: 10.1016/j.arth.2007.10.022. Epub 2008 Oct 25. PMID 18951761
- [Background] Chalidis BE, Sachinis NP, Papadopoulos P, Petsatodis E, Christodoulou AG, Petsatodis G. Long-term results of posterior-cruciate-retaining Genesis I total knee arthroplasty. J Orthop Sci. 2011 Nov;16(6):726-31. doi: 10.1007/s00776-011-0152-1. Epub 2011 Sep 10. PMID 21909722
- [Background] Kim YH, Choi Y, Kwon OR, Kim JS. Functional outcome and range of motion of high-flexion posterior cruciate-retaining and high-flexion posterior cruciate-substituting total knee prostheses. A prospective, randomized study. J Bone Joint Surg Am. 2009 Apr;91(4):753-60. doi: 10.2106/JBJS.H.00805. PMID 19339558